CLINICAL TRIAL: NCT02824315
Title: A Phase 1, Open-label, Fixed Sequence Study to Investigate the Pharmacokinetic Interaction Between 2 Direct Acting Antiviral Agents Odalasvir and AL-335 and Between 3 Direct Acting Antiviral Agents Simeprevir, Odalasvir and AL-335 at Steady State in Healthy Japanese Subjects
Brief Title: Study to Investigate the Pharmacokinetic Interaction Between 2 Direct Acting Antiviral Agents Odalasvir and AL-335 and Between 3 Direct Acting Antiviral Agents Simeprevir, Odalasvir and AL-335 at Steady State in Healthy Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108179; 64294178HPC1006 (Other: Janssen Research & Development, LLC); 2016-000950-36 (EudraCT Number)
Record Dates: First submitted 2016-06-07; First posted 2016-07-06 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — adafosbuvir; odalasvir; Simeprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AL-335+Simeprevir (SMV)+Odalasvir (ODV) (Experimental): Participants will receive AL-335 800 milligram (mg) once daily from day 1-3; SMV 75 mg once daily from Day 4-13; loading dose of ODV 150 mg on Day 14, followed by ODV 50 mg once daily from Day 15 to 23; ODV 50 mg once daily + AL-335 800 mg once daily from day 24-26; ODV 50 mg once daily + SMV 75 mg once daily from Day 27-33 and ODV 50 mg once daily + SMV 75 mg once daily + AL-335 800 mg once daily from Day 34 to 36.
  Interventions: Drug: AL-335; Drug: Odalasvir (ODV); Drug: Simeprevir (SMV)

INTERVENTIONS:
Drug: AL-335 — AL--335 800 mg once daily on Days 1--3, 24--26 and 34--36.
Drug: Odalasvir (ODV) — ODV 150 mg on Day 14 and 50 mg once daily on Days 15--23, 24--26, 27--33 and 34--36.
Drug: Simeprevir (SMV) — Simeprevir 75 mg once daily on Days 4-13, 27--33 and 34--36.

SUMMARY:
The purpose of this study is to investigate the steady-state pharmacokinetics (PK) of simeprevir (SMV), odalasvir (ODV) and AL-335 (and its metabolites ALS-022399 and ALS 022227), when these drugs are co-administered in healthy Japanese participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be a Japanese participant who has resided outside Japan for no more than 5 years and whose parents and grandparents are Japanese as determined by participant's verbal report
* Participant must have a body mass index (BMI: weight in kilogram (kg) divided by the square of height in meters) of 18.0 to 30.0 kilogram per meter square (kg/m^2), extremes included, and a body weight not less than 50.0 kg
* Participant must be healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at Screening. If there are abnormalities, the participant may be included only if the Investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the Investigator
* Participant must have a blood pressure (after the participant is supine for 5 minutes) between 90 and 140 milligram of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic. If blood pressure is out of range, up to 2 repeated assessments are permitted
* Female participant must agree to not donate eggs (ova, oocytes) for the purpose of assisted reproduction during the study and for a period of 60 days after last study drug administration or until the last follow-up visit, whichever occurs later

Exclusion Criteria:

* Participant has a history of liver or renal insufficiency (estimated creatinine clearance below 80 milliliters per minute [mL/min]); significant cardiac, vascular, pulmonary, gastrointestinal (such as significant diarrhea, gastric stasis, or constipation that in the Investigator's opinion could influence drug absorption or bioavailability), endocrine, neurologic, hematologic, rheumatologic, psychiatric, neoplastic, or metabolic disturbances
* Participant with a past history of heart arrhythmias (example- extra systolic beats or tachycardia at rest); risk factors associated with Torsade de Pointes such as hypokalemia or family history of short/long QT syndrome or sudden unexplained death (including sudden infant death syndrome) in a first degree relative [example- sibling, offspring, or biological parent])
* Participant with any history of clinically significant skin disease such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, or urticaria
* Participant has known allergies, hypersensitivity, or intolerance to simeprevir (SMV), odalasvir (ODV), AL-335 or their excipients
* Participant is a woman who is pregnant, or breast-feeding, or planning to become pregnant from signing of Informed Consent Form (ICF) until 60 days after last study drug administration or until the last follow-up visit, whichever occurs later

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2016-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Average Analyte Concentration at Steady State (Cavg,ss) | Up to Day 36
  The Cavg,ss is calculated as area under the plasma concentration-time curve during a dosing Interval (AUC[tau]) divided by the dosing interval (tau).
Maximum Observed Analyte Concentration (Cmax) | Up to Day 36
  The Cmax is the maximum observed analyte concentration.
Minimum Observed Analyte Concentration (Cmin) | Up to Day 36
  The Cmin is the minimum observed analyte concentration during dosing interval.
Trough Plasma Concentration (Ctrough) | Up to Day 36
  The (Ctrough) is the plasma concentration before dosing or at the end of the dosing interval of any dose other than the first dose in a multiple dosing regimen.
Time to Reach Maximum Observed Analyte Concentration (Tmax) | Up to Day 36
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Area Under the Analyte Concentration-Time Curve From Time 0 to 24 Hours (AUC24) | Up to Day 36
  The AUC24 is the area under the analyte concentration-time curve from time 0 to 24 hours.
Fluctuation Index (FI) | Up to Day 36
  Fluctuation Index is defined as percentage of fluctuation (variation between maximum and minimum concentration at steady state), calculated as: 100*([Cmax-Cmin]/Cavg).
Area Under the Analyte Concentration-Time Curve From Time Zero to Time of the Last Quantifiable Concentration (AUClast) | Up to Day 36
  The (AUC [0-last]) is the area under the analyte concentration-time curve from time 0 to time of the last quantifiable concentration.
Area Under the Analyte Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) | Up to Day 36
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Elimination Rate Constant (Lambda[z]) | Up to Day 36
  Lambda(z) is first-order elimination rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Elimination Half-Life (t1/2) | Up to Day 36
  Elimination half-life (t[1/2]) is associated with the terminal slope (lambda [z]) of the semi-logarithmic drug concentration-time curve, calculated as 0.693/lambda(z).

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AE) as a Measure of Safety and Tolerability | Up to Follow-up (170 to 175 days after last study drug intake)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Surrey, United Kingdom